CLINICAL TRIAL: NCT06668571
Title: Central and Peripheral GABA and Glutamate Modulation With Intravenous Ketamine for Treatment-Resistant Depression (G2K): A Randomized, Double-Blind, Placebo-Controlled Study
Brief Title: Intravenous Ketamine for Treatment-Resistant Depression
Acronym: G2K
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Balwinder Singh, MD, MS, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 24-005249; 5KL2TR002379 (NIH); 5KL2TR002379-08 (NIH)
Record Dates: First submitted 2024-10-16; First posted 2024-10-31 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Depressive Disorder, Treatment-Resistant; Treatment Resistant Depression (TRD)
Keywords: Major Depression; Depressive Disorder, Treatment-Resistant; MDD; TRD; Treatment-Resistant Depression; Treatment-Resistant Major Depression; Ketamine; Intravenous Ketamine
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major | interventions — Ketamine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: MRI-tech, Radiologist, and Clinical Research Trial Unit Nurses. Any staff involved in the ratings will be blinded to the treatment of the subject for infusion. Only the study investigator present during infusion in the MRI will be unblinded for safety precautions during the infusion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine Group (Experimental): Subjects will receive IV racemic ketamine at a dose of 0.5 mg per kg of the participant's actual body weight, with a maximum dose of 50 mg for individuals weighing over 100 kg.
  Interventions: Drug: Ketamine
- Normal Saline/Placebo Group (Placebo Comparator): Subjects will receive an IV infusion of normal saline over a duration of 40 minutes
  Interventions: Drug: Normal Saline

INTERVENTIONS:
Drug: Ketamine — The subjects will receive 1:1 single IV racemic ketamine (dosed @0.5 mg/kg actual body weight) (n=15) 40-min infusion in an MRI scanner, followed by an optional open-label ketamine infusion (available to everyone) 1-7 days after the initial treatment
  Arms: Ketamine Group
Drug: Normal Saline — The subjects will receive 1:1 single IV normal saline/placebo (n=15) 40-min infusion in an MRI scanner, followed by an optional open-label ketamine infusion (available to everyone) 1-7 days after the initial treatment
  Arms: Normal Saline/Placebo Group

SUMMARY:
The purpose of this study is to to evaluate the relationships between peak (% change from baseline) central GABA and Glu levels during a 40-min IV ketamine or normal saline infusion utilizing fMRS, and change in peripheral GABA and Glu levels from baseline to 24-hr postinfusion utilizing LCMS, with baseline to 24-hr post-infusion change in depression (MADRS) in 30 TRD adults.

DETAILED DESCRIPTION:
This will be a randomized, double-blind, placebo-controlled, parallel-group study where adult subjects with treatment refractory major depressive disorder (MDD) will receive 1:1 single IV racemic ketamine (n=15) or normal saline (placebo) (n=15) infusion in an MRI scanner, followed by an optional open-label ketamine infusion. In this innovative comparative study utilizing novel dynamic sliding-window fMRS and liquid chromatography-mass spectrometry (LCMS), we will investigate the dynamic relationship between GABA and Glu levels measured centrally and peripherally, respectively, with change in depression symptoms utilizing the Montgomery Asberg Depression Rating Scale (MADRS).12 Given preclinical models of reduced ACs and glutamatergic function in depression, we will also include an exploratory analysis of ACs metabolomic markers associated with ketamine treatment response.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* Meets diagnostic criteria for major depressive disorder without psychotic features per the SCID DSM-IV-TR
* PHQ-9 total score ≥ 15 at screening
* Treatment-resistant depression, as defined by failure of at least two previous antidepressant treatments within the current depressive episode. Failed antidepressant treatments can include pharmacotherapy for depression at an adequate dose for at least 8 weeks, trial of transcranial magnetic stimulation (TMS) or an acute series of at least 6 administrations of electroconvulsive therapy (ECT)
* Ability to pass a comprehension assessment test related to effects of ketamine and trial objectives and criteria

Exclusion Criteria:

* Inability to speak English
* Inability to provide consent or have a legal guardian
* Patients with a BMI > 40 kg/m2.
* Personality disorder being the primary diagnosis
* Diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or active psychotic symptoms
* Active post-traumatic stress disorder symptoms based on clinical assessment
* Ongoing prescription of > 2 mg lorazepam equivalents (total) daily, or morning dosing of any benzodiazepine at the time of assessment
* Medications known to affect glutamate (i.e., Riluzole, Carbamazepine) or GABA (zaleplon, zolpidem, zopiclone, Valproate, Gabapentin, Pregabalin, tiagabine, and vigabatrin) are prohibited within two weeks prior to administration of study drug and at least 24 hours after last dose of study drug
* Monoamine Oxidase Inhibitors (MAOIs) are prohibited two weeks prior to administration of study drug
* Opioid antagonists (naltrexone, naloxone, nalmefene, methylnaltrexone, buprenorphine and naloxone combination) are prohibited within two weeks prior to administration of study drug and at least 24 hours after last dose of study drug
* CYP3A4 inducers carbamazepine and modafinil are prohibited within two weeks prior to administration of study drug and at least 24 hours after last dose of study drug.
* Currently undergoing TMS, vagal nerve stimulation, or deep brain stimulation as either an acute or maintenance treatment of depression
* ECT in the past 6 months
* Any active or unstable medical condition judged by the study psychiatrist as conferring too great a level of medical risk to allow inclusion in the study
* A history of bleeding in the brain
* Arteriovenous malformation or a history of aneurysm
* Use of methamphetamine, cocaine, or cannabis. Abuse of stimulant (s) within the prior 12 months
* Any current substance use disorder (excluding nicotine and caffeine). Note: Persons will be allowed to enroll in this study if their substance use is in complete (not partial) and sustained (> 1 year) remission
* History of traumatic brain injury that resulted in loss of consciousness with brain bleeding
* History of tonic-clonic (grand mal) seizures
* Developmental delay, intellectual disability, or intellectual disorder
* Clinical or self-reported diagnosis of delirium, encephalopathy, or related clinical diagnosis within the prior 12 months
* Minor or Major Neurocognitive disorder
* Received ketamine treatment for depression within the prior 2 months
* History of either poor antidepressive response to or poor tolerability of ketamine (any route of administration) when previously administered
* History of hypothyroidism unless taking a stable dose of thyroid medication and asymptomatic for 3 months
* Hepatic insufficiency (2.5 X ULN for AST or ALT) within 3 months of consent, past liver transplant recipient, and/or clinical diagnosis of cirrhosis of the liver
* Gastroesophageal reflux disease that is poorly managed
* A diagnosis of Complex Regional Pain Syndrome (CRPS)
* Pregnancy, or nursing
* History of claustrophobia with active symptoms that would interfere with the MRI
* Any contraindication to MRI safety questionnaire
* Poorly controlled hypertension.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Peak (% change from baseline) Anterior Cingulate Cortex metabolites (Gamma-Aminobutyric Acid and Glutamate) | Baseline to the end of 40-minute infusion
  To measure peak (% change from baseline) Anterior Cingulate Cortex (ACC) Gamma-Aminobutyric Acid (GABA) and Glutamate (Glu) levels during a 40-minute IV ketamine or normal saline (0.9% sodium chloride) infusion utilizing fMRS (functional Magnetic Resonance Spectroscopy)
Change in peripheral Gamma-Aminobutyric Acid and Glutamate levels | Baseline to the end of 40-minute infusion
  Change in peripheral Gamma-Aminobutyric Acid (GABA) and Glutamate (Glu) levels measured utilizing liquid chromatography-mass spectrometry (LCMS) at baseline and the end of 40-minute infusion
Change in the Montgomery Asberg Depression Rating Scale | Baseline to 24-hours post-infusion
  Montgomery Asberg Depression Rating Scale (MADRS) is a 10-item clinician rating of depressive symptoms used in the previous ketamine research studies. Higher scores represent higher levels of depression.
Correlation between the percent change in central (anterior cingulate cortex) Gamma-Aminobutyric Acid and Glutamate levels and the change in depression severity measured using the Montgomery-Åsberg Depression Rating Scale | Baseline to the end of 40-minute infusion for GABA and Glu. Baseline to 24 hours post-infusion for MADRS
  Outcome measure: Changes in the total Montgomery-Asberg Depression Rating Scale (MADRS) scale from baseline (pre-infusion) to 24 hours post-infusion. MADRS will be compared by randomized arm as a continuous variable as well as defined by remission status (MADRS≤9). The total MADRS score can range from 0 to 60, with higher scores indicating a worse outcome.
  We aim to evaluate the correlation between the percent change in anterior cingulate cortex (ACC) Gamma-Aminobutyric Acid (GABA) and Glutamate (Glu) levels (from baseline to peak) during a 40-minute IV infusion of ketamine or normal saline (0.9% sodium chloride) using functional magnetic resonance spectroscopy (fMRS) and the change in MADRS scores (from baseline to 24 hours).
Correlation between the percent change in serum Gamma-Aminobutyric Acid and Glutamate levels and the change in depression severity measured using the Montgomery-Åsberg Depression Rating Scale | Baseline to the end of 40-minute infusion for serum GABA and Glu. Baseline to 24 hours post-infusion for MADRS
  Outcome measure: Changes in the total Montgomery-Asberg Depression Rating Scale (MADRS) scale from baseline (pre-infusion) to 24 hours post-infusion. MADRS scores will be compared by randomized arm as a continuous variable as well as defined by remission status (MADRS≤9). The total MADRS score can range from 0 to 60, with higher scores indicating a worse outcome.
  We aim to evaluate the correlation between the percent change in serum Gamma-Aminobutyric Acid (GABA) and Glutamate (Glu) levels during a 40-minute IV infusion of ketamine or normal saline (0.9% sodium chloride) using Liquid Chromatography-Mass Spectrometry (LCMS) and the change in MADRS scores (from baseline to 24 hours).

SECONDARY OUTCOMES:
Change in McIntyre And Rosenblat Rapid Response Scale | Baseline to up to 24 hours post-infusion
  The McIntyre and Rosenblat Rapid Response Scale (MARRRS) is a validated self-report instrument designed to assess rapid treatment response in the context of rapid-acting antidepressant drugs (RAADs), such as ketamine. The scale comprises 14 items and has shown promising psychometric properties, including high internal consistency and significant convergent validity. Each item is scored on a 4-point ordinal scale, where 0 indicates the absence of symptoms and 3 signifies the highest severity of symptoms. The total score ranges from 0 to 42, with higher scores indicating a more severe state of depression.
Change in Quick Inventory of Depressive Symptomatology (Self-Report) | Baseline to up to 24 hours post-infusion
  The Quick Inventory of Depressive Symptomatology (QIDS-SR-16) is a depression scale that assesses the symptom domains of major depressive disorder, with scores ranging from 0 to 27. Higher scores indicate more severe depressive symptoms. The individual items evaluate key aspects such as sadness, anhedonia (the loss of pleasure), and sleep disturbances, which may manifest as insomnia or hypersomnia. Additionally, the scale addresses changes in appetite or weight and includes assessments of psychomotor agitation or retardation. It also measures fatigue or loss of energy, feelings of worthlessness or excessive guilt, and difficulties in concentration. Furthermore, the scale incorporates items related to suicidal ideation, offering a comprehensive overview of both the emotional and physical symptoms experienced by individuals with depression.
Changes in short chain acylcarnitine levels | Baseline to up to 24 hours post-infusion.
  Changes in short-chain acylcarnitine (AC) levels-early change (baseline to 40 minutes) and late change (100 minutes to 24 hours)-among patients who received a 40-minute IV infusion of either ketamine or normal saline (0.9% sodium chloride).
Changes in short-chain acylcarnitine levels and ketamine-related remission | Baseline to up to 24 hours post-infusion.
  To evaluate the relationship between changes in short-chain AC levels-early change (baseline to 40 minutes) and late change (100 minutes to 24 hours)-among remitters and non-remitters (MADRS < 10) at 24 hours.
Changes in mTOR (mechanistic Target of Rapamycin) | Baseline to the end of 40-minute infusion
  To investigate the changes in mTOR from baseline to the end of infusion with IV ketamine compared to normal saline. To investigate the correlation between anhedonia phenotypes (baseline) and the percent change in mTOR from baseline. Anhedonia phenotypes will be assessed using the MADRS and the SHAPS.
Change in the Snaith-Hamilton Pleasure Scale | Baseline to up to 24 hours post-infusion
  The Snaith-Hamilton Pleasure Scale (SHAPS) is a 14-item scale that measures anhedonia, the inability to experience pleasure. The items cover the domains of: social interaction, food and drink, sensory experience, and interest/pastimes. A score of 2 or less constitutes a "normal" score, while an "abnormal" score is defined as 3 or more. A higher total score indicates greater levels of anhedonia.
Changes in neurocognitive functioning | Baseline to 24 hours post-infusion
  The Repeatable Battery for the Assessment of Neuropsychological Status (RBANS)is a brief, standardized, individually administered battery to measure cognitive change in immediate memory, visuospatial/constructional orientation, language (naming, fluency), attention, and delayed memory. The 12 subtests that comprise the RBANS require approximately 30 minutes to administer.
Change in Beck Scale for Suicidal Ideation | Baseline to up to 24 hours post-infusion
  The Beck Scale for Suicidal Ideation consists of 19 items which can be used to evaluate a patient's suicidal intentions. It can also be used to monitor a patient's response to interventions over time. Each of the 19 items is rated on a 0-3 point scale (range 0-38, with higher scores indicating greater suicidal ideations or risk), and includes specific items that assess wish to live, wish to die, desire to make an active suicide attempt, passive suicidal desire, duration of suicidal ideations, frequency of suicidal ideations, and subjective level of control over suicidal actions.
Changes in Dimensional Anhedonia Rating Scale | Baseline to up to 24 hours post-infusion
  The Dimensional Anhedonia Rating Scale (DARS) measures anhedonia, including facets of desire, motivation, effort, and consummatory pleasure. The scale has demonstrated high internal consistency, reliability, and validity across studies. It has shown superiority in distinguishing MDD subgroups. The DARS total score ranges from 0 to 68. A lower DARS score reflects more severe anhedonia, while a higher score indicates lower anhedonia.
Change in Clinical Global Impression | Baseline to up to 24 hours post-infusion
  The Clinical Global Impression (CGI) is assessed using a 7-point scale. The CGI-Severity (CGI-S) of Illness measures the severity of the patient's condition, ranging from 1 (normal) to 7 (among the most severely ill patients). In addition, the CGI-Improvement (CGI-I) scale evaluates changes in the patient's condition from baseline, which is prior to the ketamine infusion. The CGI-I scale is rated as follows: 1 indicates "very much improved" since the initiation of treatment, 2 signifies "much improved," 3 denotes "minimally improved," 4 represents "no change from baseline," 5 means "minimally worse," 6 indicates "much worse," and 7 reflects "very much worse" since the initiation of treatment.
Perceived Stress | Baseline to up to 24 hours post-infusion
  The Perceived Stress Scale is a 10-item self-rated tool that measures the frequency of an individual's perception of stress over the last month
Resilience | Baseline to 24 hours post-infusion
  The Brief Resilience Scale (BRS) is a reliable tool for assessing resilience, specifically focused on an individual's ability to bounce back or recover from stress. The BRS ranges from 1 to 5, with higher scores indicating greater resilience-that is, a stronger ability to bounce back from stress.

CONTACTS AND LOCATIONS:
Overall Officials: Balwinder Singh, M.D., M.S., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: Yes
The study results will be uploaded to the website after the completion of the study. All related research findings will be published or submitted to the NIH.
Time Frame: 2027
Access Criteria: The study results will be uploaded to the website after the completion of the study.

REFERENCES:
- [Background] Singh B, Vande Voort JL, Pazdernik VK, Frye MA, Kung S. Treatment-resistant depression patients with baseline suicidal ideation required more treatments to achieve therapeutic response with ketamine/esketamine. J Affect Disord. 2024 Apr 15;351:534-540. doi: 10.1016/j.jad.2024.01.262. Epub 2024 Jan 30. PMID 38302067
- [Background] Singh B, Bobo WV, Rasmussen KG, Stoppel CJ, Rico JA Jr, Schak KM, Biernacka JM, Frye MA, Vande Voort JL. The Association Between Body Mass Index and Remission Rates in Patients With Treatment-Resistant Depression Who Received Intravenous Ketamine. J Clin Psychiatry. 2019 Nov 12;80(6):19l12852. doi: 10.4088/JCP.19l12852. No abstract available. PMID 31721482
- [Background] Frye MA, Blier P, Tye SJ. Concomitant benzodiazepine use attenuates ketamine response: implications for large scale study design and clinical development. J Clin Psychopharmacol. 2015 Jun;35(3):334-6. doi: 10.1097/JCP.0000000000000316. No abstract available. PMID 25928701
- [Background] Singh B, Parikh SV, Voort JLV, Pazdernik VK, Achtyes ED, Goes FS, Yocum AK, Nykamp L, Becerra A, Smart L, Greden JF, Bobo WV, Frye MA, Burdick KE, Ryan KA. Change in neurocognitive functioning in patients with treatment-resistant depression with serial intravenous ketamine infusions: The Bio-K multicenter trial. Psychiatry Res. 2024 May;335:115829. doi: 10.1016/j.psychres.2024.115829. Epub 2024 Feb 28. PMID 38479192
- [Background] Parikh SV, Vande Voort JL, Yocum AK, Achtyes E, Goes FS, Nykamp L, Singh B, Lopez-Vives D, Sera CE, Maixner D, Tarnal V, Severe J, Bartek S, Tye SJ, Rico J, Stoppel CJ, Becerra A, Smart L, Miller CR, Frye MA, Greden JF, Bobo WV. Clinical outcomes in the biomarkers of ketamine (Bio-K) study of open-label IV ketamine for refractory depression. J Affect Disord. 2024 Mar 1;348:143-151. doi: 10.1016/j.jad.2023.12.033. Epub 2023 Dec 22. PMID 38142892
- [Background] Singh B, Kung S, Pazdernik V, Schak KM, Geske J, Schulte PJ, Frye MA, Vande Voort JL. Comparative Effectiveness of Intravenous Ketamine and Intranasal Esketamine in Clinical Practice Among Patients With Treatment-Refractory Depression: An Observational Study. J Clin Psychiatry. 2023 Feb 1;84(2):22m14548. doi: 10.4088/JCP.22m14548. PMID 36724113
- [Background] Vande Voort JL, Morgan RJ, Kung S, Rasmussen KG, Rico J, Palmer BA, Schak KM, Tye SJ, Ritter MJ, Frye MA, Bobo WV. Continuation phase intravenous ketamine in adults with treatment-resistant depression. J Affect Disord. 2016 Dec;206:300-304. doi: 10.1016/j.jad.2016.09.008. Epub 2016 Sep 12. PMID 27656788
- [Background] Brix MK, Ersland L, Hugdahl K, Dwyer GE, Gruner R, Noeske R, Beyer MK, Craven AR. Within- and between-session reproducibility of GABA measurements with MR spectroscopy. J Magn Reson Imaging. 2017 Aug;46(2):421-430. doi: 10.1002/jmri.25588. Epub 2017 Feb 15. PMID 28205280
- [Background] Dubin MJ, Mao X, Banerjee S, Goodman Z, Lapidus KA, Kang G, Liston C, Shungu DC. Elevated prefrontal cortex GABA in patients with major depressive disorder after TMS treatment measured with proton magnetic resonance spectroscopy. J Psychiatry Neurosci. 2016 Apr;41(3):E37-45. doi: 10.1503/jpn.150223. PMID 26900793
- [Background] Port JD, Singh B, Frye MA. Dynamic Sliding-Window MRS Method for Measuring Changes in Glutamate and GABA in Patients with Major Depressive Disorder. presented at: ISMRM & SMRT Virtual Conference & Exhibition; 2020; Virtual https://www.ismrm.org/20/program_files/DP01-09.htm#044
- [Background] Singh B, Vande Voort JL, Riva-Posse P, Pazdernik VM, Frye MA, Tye SJ. Ketamine-Associated Change in Anhedonia and mTOR Expression in Treatment-Resistant Depression. Biol Psychiatry. 2023 Jun 15;93(12):e65-e68. doi: 10.1016/j.biopsych.2022.10.007. Epub 2023 Jan 25. No abstract available. PMID 36707268
- [Background] Rotroff DM, Corum DG, Motsinger-Reif A, Fiehn O, Bottrel N, Drevets WC, Singh J, Salvadore G, Kaddurah-Daouk R. Metabolomic signatures of drug response phenotypes for ketamine and esketamine in subjects with refractory major depressive disorder: new mechanistic insights for rapid acting antidepressants. Transl Psychiatry. 2016 Sep 20;6(9):e894. doi: 10.1038/tp.2016.145. PMID 27648916
- [Background] Singh B, Port JD, Voort JLV, Coombes BJ, Geske JR, Lanza IR, Morgan RJ, Frye MA. A preliminary study of the association of increased anterior cingulate gamma-aminobutyric acid with remission of depression after ketamine administration. Psychiatry Res. 2021 Jul;301:113953. doi: 10.1016/j.psychres.2021.113953. Epub 2021 Apr 20. PMID 33933839
- [Background] Singh B, Port JD, Pazdernik V, Coombes BJ, Vande Voort JL, Frye MA. Racemic ketamine treatment attenuates anterior cingulate cortex GABA deficits among remitters in treatment-resistant depression: A pilot study. Psychiatry Res Neuroimaging. 2022 Mar;320:111432. doi: 10.1016/j.pscychresns.2021.111432. Epub 2021 Dec 24. No abstract available. PMID 34973601
- [Background] Singh B, MahmoudianDehkordi S, Voort JLV, Han X, Port JD, Frye MA, Kaddurah-Daouk R; Mood Disorders Precision Medicine Consortium (MDPMC). Metabolomic signatures of intravenous racemic ketamine associated remission in treatment-resistant depression: A pilot hypothesis generating study. Psychiatry Res. 2022 Aug;314:114655. doi: 10.1016/j.psychres.2022.114655. Epub 2022 May 28. PMID 35738038